CLINICAL TRIAL: NCT05428280
Title: Effectiveness of Muscle Energy Technique Versus Myofascial Mobilization in Improving Functional Outcome in Sub-acute Non-specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Comparing the Effects of Muscle Energy Technique Versus Myofascial Mobilization in Managing Sub-acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Faizan Abdullah, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAbdullah
Record Dates: First submitted 2022-06-13; First posted 2022-06-23 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Lordosis; Low Back Pain
MeSH Terms: conditions — Lordosis; Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Techniques (Experimental): Following physiotherapy will be given to the participants in this group for 4 weeks, 3 times a week:
  1. Muscle Energy Technique
  Interventions: Other: Physiotherapy; Other: Muscle Energy technique
- Myofascial Mobilization Techniques (Active Comparator): Following physiotherapy will be given to the participants in this group for 4 weeks, 3 times a week:
  1. Myofascial Mobilization
  Interventions: Other: Physiotherapy; Other: Myofacial mobilization

INTERVENTIONS:
Other: Physiotherapy — Conventional treatment consisted of Transcutaneous Electrical Nerve Stimulation and Progressive Back Strengthening Exercise
Other: Muscle Energy technique — Muscle Energy Technique (MET) is a technique that was developed in 1948 by Fred Mitchell, Sr, D.O[1]. It is a form of manual therapy, widely used in Osteopathy, that uses a muscle's own energy in the form of gentle isometric contractions to relax the muscles via autogenic or reciprocal inhibition and lengthen the muscle.
  Arms: Muscle Energy Techniques
Other: Myofacial mobilization — It is a type of gentle, constant massage that releases tightness and pain throughout your myofascial tissues
  Arms: Myofascial Mobilization Techniques

SUMMARY:
Institute for Clinical Systems Improvement (ICSI) defines sub-acute low back pain as low back pain lasting between 4 and 12 weeks. There is insufficient evidence regarding the comparative effect of muscle energy technique and myofascial mobilization in the management of sub-acute non-specific low back pain with the tightness of quadratus lumborum and erector spinae muscles

DETAILED DESCRIPTION:
A randomized experimental controlled trial will be carried out to compare the effectiveness of muscle energy technique and myofascial mobilization in the management of sub-acute non-specific low back pain. A total of 60 male and female volunteers having subjects with sub-acute nonspecific low back pain will be recruited in this study. Subjects will be assessed at baseline for pain and disability using Visual Analogue Scale and Ronald Morris Disability Questionnaire (RMDQ 0-24) respectively. After baseline assessment, all subjects will be allocated to two groups through computer-generated random sampling. Group 1 will perform Muscle energy technique combined with conventional exercise; Group 2 will receive Myofascial Mobilization combined with conventional exercise. This study will be conducted at the Physiotherapy Department of Sindh Institute of Physical Medicine and Rehabilitation (SIPM&R). Data will be analyzed using SPSS 21 and ANCOVA technique will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute low back pain with the range of 7 to 12 weeks of unresolved symptoms.
* Positive test of tight Erector spinae muscle and Tight Quadratus Lumboram muscle

Exclusion Criteria:

* Spinal malignancy
* Spinal fracture
* Spine foraminal stenosis
* Nerve root compression
* Radicular symptoms
* Sciatica
* Cord compression
* Paralysis
* Muscular dystrophy
* Myelopathy
* Seizure disorder
* Severe trauma
* Unexplained weight loss

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Change from baseline pain intensity at 4 weeks
  The visual analogue scale is used for measurement of pain intensity. It is a continuous scale. It comprises a horizontal or vertical 10 centimeters or 100 millimeters line. The participant is asked to indicate a point of pain intensity by placing a line perpendicular to the Visual analogue scale line. The scale is most commonly referred by "no pain" with score of 0 and "worst imaginable pain" with score of 100 on the scale. The higher scores shows higher pain intensity and lower scores shows lower pain intensity.
Rolland Morris Disability Questionnaire | Change from baseline functional disability at 4 weeks
  It is a standard questionnaire with questions regarding pain and the disabling effect on daily activities. Its score ranges from 0 to 24 (no disability to maximum disability)

CONTACTS AND LOCATIONS:
Overall Officials: Faizan Abdullah, MSAPT, DPT, Principal Investigator — Sindh Institute of Physical Medicine and Rehabilitation
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No